CLINICAL TRIAL: NCT02149836
Title: A Proof-Of-Concept Clinical Trial of a Novel KCNQ Potentiator in Major Depressive Disorder
Brief Title: Study to Treat Major Depressive Disorder (MDD) With a New Medication
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, James Murrough, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 14-0597
Record Dates: First submitted 2014-05-22; First posted 2014-05-29 (Estimated); Results first posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-03

CONDITIONS: Major Depressive Disorder; Depression
Keywords: major depressive disorder; depression; treatment resistent depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — ezogabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ezogabine (Experimental): Ezogabine dosage plan to 900mg and then tapered down
  Interventions: Drug: ezogabine

INTERVENTIONS:
Drug: ezogabine — Treatment Week 1: 100mg of Ezogabine by mouth three times per day (total daily dose = 300mg) Treatment Week 2: dose will be increased to 150 mg Ezogabine by mouth three times per day (total daily dose = 450mg).
  Treatment Week 3: dose will be increased to 200mg of Ezogabine by mouth three times per day (total daily dose = 600mg).
  Treatment Week 4: dose will be increased to 250mg of Ezogabine by mouth three times per day (total daily dose = 750mg).
  Treatment Week 5: dose will be increased to 300mg of Ezogabine by mouth three times per (total daily dose = 900mg).
  Participants will continue to take 900mg of Ezogabine per day and return weekly to the clinic for the remainder of the study.
  Following this primary outcome visit, participants will be instructed to taper the study medication over the following 3 weeks based on FDA recommended guidelines as follows:
  250 mg po TID daily x 1 week, then 200 mg po daily x 1 week, then 100 mg po daily x 1 week, then discontinue
  Other Names: Potiga; Retigabine

SUMMARY:
The purpose of this study is to test the antidepressant effects of Ezogabine in major depressive disorder (MDD). The investigators also aim to determine the safety and tolerability Ezogabine in patients with MDD. The investigators hypothesize that depressive symptoms will be significantly decreased following an 8-week treatment period of the medication compared to baseline.

DETAILED DESCRIPTION:
Study Introduction:

Major depressive disorder (MDD) is a global health disease associated with significant morbidity and costs. Many anti-depressants exist within the monoaminergic system yet novel therapeutics are still needed outside of this system. Ezogabine, currently approved by the FDA for adjunctive treatment of partial-onset seizures, may serve as a potential key agent for those with MDD. Ezogabine is known to bind to and activate KCNQ transmembrane K+ ion channels, specifically targeting KCNQ2 in the VTA. Such membrane activity has been show to play a role in previous studies involving a social defeat model of depression. Specifically, data has shown that KCNQ channels were upregulated only in resilient mice and moreover, ezogabine was able to potentiate KCNQ channel activity to result in a fast reversal of the depressed phenotype.

General Investigational Plan:

Objectives:

A. Primary Efficacy Objective: To test the antidepressant effects of Ezogabine in MDD.

B. Primary Safety Objective: To characterize the safety and tolerability of Ezogabine in patients with MDD.

C. Secondary Objectives: To measure the effects of Ezogabine on ventral tegmental area (VTA)-striatal reward circuitry in MDD using reward task-based functional MRI. Rationale: Ezogabine is hypothesized to modulate the firing rate of VTA dopamine (DA) neurons and thereby influence the functioning of the mesolimbic reward system.

Hypotheses

A. Efficacy Hypothesis:

Hypothesis 1a: Depressive symptoms will be significantly decreased following an 8-week treatment period compared to baseline, as measured by change in Montgomery-Åsberg Depression Rating Scale (MADRS).

Hypothesis 1b: The antidepressant response rate at study end (defined as 50% in depressive symptoms compared to baseline) will exceed 50%, consistent with known response rates of current antidepressant agents.

B. Safety Hypothesis: Ezogabine will be safe and adverse event rates will be similar to rates observed in other adult populations. Specific safety items to be monitored include frequency and intensity of adverse events as measured by the Patient Rated Inventory of Side Effects (PRISE) and treatment-emergent suicidal ideation or behavior as measured by the Columbia-Suicide Severity Rating Scale (C-SSRS).

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants, 18-65 years of age;
* Current diagnosis of major depressive disorder according as determined by a psychiatrist and confirmed with The Mini-International Neuropsychiatric Interview (MINI);
* At least moderate depression severity as defined by a score of >= 21 on the Montgomery-Asberg Depression Rating Scale (MADRS);
* At least a moderate level of anhedonia based on a Snaith-Hamilton Pleasure Scale (SHAPS) score ≥ 20;
* If female of childbearing potential, must agree to use of a medically accepted form of contraception, or else agree to abstinent;
* Participants must have a level of understanding of the English language sufficient to agree to all tests and examinations required by the study and must be able to participate fully in the informed consent process.

Exclusion Criteria:

* Lifetime diagnosis of schizophrenia or any psychotic disorder, bipolar disorder, obsessive compulsive disorder or pervasive developmental disorders or mental retardation;
* Diagnosis of a substance use disorder within the past 6 months (excluding substance use disorder in sustained remission)
* Female participants who are pregnant, nursing, for may become pregnant;
* Any unstable medical illnesses including hepatic, renal, gastroenterologic, respiratory, cardiovascular (including ischemic heart disease); endocrinologic, neurologic (including history of severe head injury), immunologic, or hematologic disease;
* Clinically significant abnormalities of laboratories, physical examination, or ECG;
* Prolonged QT Interval at screening, operationalized as a QTc of > 480 ms at baseline;
* Hypokalemia (potassium value less than 3.5mEq/L) or hypomagnesemia (magnesium value less than 1.6mEq/L) at baseline;
* A history of retinal abnormalities (ie, pigment changes, retinal dystrophy) or findings of retinal pathology on ophthalmological exam at baseline
* Antidepressant medication within 2 weeks of start of treatment (4 weeks for fluoxetine)*
* Other psychotropic medication, including antipsychotics and mood stabilizers within 2 weeks of start of treatment; subjects will be allowed to remain on a stable dose of zolpidem 10 mg nightly for sleep or a benzodiazepine as needed for sleep or anxiety (dosage equivalent to lorazepam 1 mg daily or less)
* No current or recent significantly elevated risk of self-harm or violence as determined by the PI.
* For subjects who may participate in the MRI portion of the study, claustrophobia, any trauma or surgery which may have left magnetic material in the body, magnetic implants or pacemakers, and inability to lie still for 1 hour or more.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Murrough, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Ezogabine: Ezogabine dosage plan starts at 100mg 3x/day and increased to 300mg 3x/day and then tapered down to discontinue for the end of the study.
Period: Overall Study
Arm/Group | Ezogabine
Started | 18
Completed | 17
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ezogabine
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.1 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 5
MADRS [Mean (Standard Deviation); unit: units on a scale] — The Montgomery-Asberg Depression Rating Scale (MADRS) has 10-items which are based on mood symptoms over the past 7 days. Each items is scored 0 (normal) to 6 (severe depression) with overall score ranges from 0 (normal) to 60 (severe depression).
  units on a scale | 29.50 (4.93)
QIDS [Mean (Standard Deviation); unit: units on a scale] — Quick Inventory of Depressive Symptomatology, Self-Report (QIDS-SR) score - 9-item is rated 0 to 3, with the total score range from 0 (no depression) - 27 (severe depression).
  units on a scale | 13.78 (3.19)
SHAPS [Mean (Standard Deviation); unit: units on a scale] — the Snaith-Hamilton pleasure scale - 14-item questionnaire commonly used to assess anhedonia. A total score can be derived by summing the responses to each item. Items answered with "strongly agree", or higher pleasure, are coded as "1", while a "strongly disagree", or less pleasure, response was assigned a score of "4." Total scores on the SHAPS can range from 14 to 56, with higher scores corresponding to higher levels of anhedonia.
  units on a scale | 34.28 (5.45)
TEPS-CON [Mean (Standard Deviation); unit: units on a scale] — Temporal Experience of Pleasure Scale (TEPS) - The TEPS is composed of 18-items rated on a likert-type scale ranging from 1 (Very False for me) to 6 (Very True for me), and yields two subscales measuring Anticipatory (TEPS-ANT) and Consummatory (TEPS-CON) pleasure. TEPS-CON full scale is from 9-54. Lower scores indicate greater levels of anhedonia.
  units on a scale | 21.33 (8.39)
TEPS ANT [Mean (Standard Deviation); unit: units on a scale] — Temporal Experience of Pleasure Scale (TEPS) - The TEPS is composed of 18-items rated on a likert-type scale ranging from 1 (Very False for me) to 6 (Very True for me), and yields two subscales measuring Anticipatory (TEPS-ANT) and Consummatory (TEPS-CON) pleasure. TEPS-ANT full scale is from 9-54. Lower scores indicate greater levels of anhedonia.
  units on a scale | 29.67 (4.22)
CGI-S [Mean (Standard Deviation); unit: units on a scale] — The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Considering total clinical experience, a patient is assessed on severity of mental illness at the time of rating 1, normal, not at all ill; 2, borderline mentally ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill.
  units on a scale | 4.22 (0.43)

OUTCOME MEASURES:

1. Primary Outcome: Montgomery-Asberg Depression Rating Scale Comparison to Baseline
Description: The Montgomery-Asberg Depression Rating Scale (29) is a 10-item instrument used for the evaluation of depressive symptoms in adults and for the assessment of any changes to those symptoms. Each of the 10 items is rated on a scale of 0 to 6, with differing descriptors for each item. These individual item scores are added together to form a total score, which can range between 0 and 60 points. The MADRS is specifically designed to detect changes in depression severity in the context of a medication treatment trial.
Time Frame: baseline and after end of treatment (10 weeks)
Population: 1 participant withdrew before end of study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ezogabine
Number analyzed (Participants) | 18
units on a scale
  Baseline | 29.50 (4.93)
  10 weeks: number analyzed (Participants) | 17
  10 weeks | 15.83 (7.85)

2. Secondary Outcome: Patient Rated Inventory of Side Effects (PRISE)
Description: Number of symptom events as reported by the patient in a self-report measure. PRISE assesses the presence of treatment side effects in nine organ/function systems (gastrointestinal, nervous system, heart, eyes/ears, skin, genital/urinary, sleep, sexual functioning, and other)
Time Frame: 8 weeks
Measure: Number; unit: events
Arm/Group | Ezogabine
Number analyzed (Participants) | 17
events | 105

3. Secondary Outcome: Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: The Columbia-Suicide Severity Rating Scale (C-SSRS) is a comprehensive, semi-structured interview measure that uniquely measures the full spectrum of suicidality including passive and active suicidal ideation, suicidal intent as well as suicidal behaviors. Full range from 0 (low intensity suicidal ideation to 9 (high intensity suicidal ideation).
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ezogabine
Number analyzed (Participants) | 17
units on a scale | 0.278 (0.958)

4. Secondary Outcome: Changes in Reward System Activation After Treatment With Ezogabine
Description: Functional MRI of reward processing: The primary neuroimaging endpoint is the degree of change observed in the reward system in the brain. Although it was an outcome measure, the data format is a set of 4-dimensional statistical maps and not reported in raw data. Mean changes in activation of the ventral tegmental area (VTA) or ventral striatum (VS) in response to reward cue to reward receipt, and VTA mean change in beta weight in response to reward cue at 8 weeks as compared to baseline. The Z-score indicates the number of standard deviations away from a reference population in the same age range. A Z-score of 0 is equal to the mean. Negative numbers indicate values lower than the mean and positive numbers indicate values higher than the mean.
Time Frame: baseline and post treatment (8 weeks)
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Ezogabine
Number analyzed (Participants) | 18
z-score
  VTA in response to reward cue | -0.043 (0.55)
  VTA in response to reward receipt | -0.021 (0.32)
  VS in response to reward cue | -0.031 (0.40)
  VS in response to reward receipt | 0.013 (0.23)

ADVERSE EVENTS:
Arm/Group | Ezogabine
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 15/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ezogabine (N=18)
Dizziness (Nervous system disorders) | 8
Headache (Nervous system disorders) | 2
Somnolence (Nervous system disorders) | 1
Confusional State (Nervous system disorders) | 3
Disturbance in attention (Nervous system disorders) | 1
Illusion (Psychiatric disorders) | 1
Delayed orgasm (Psychiatric disorders) | 1
Erectile Dysfunction (Psychiatric disorders) | 1
Nausea (Psychiatric disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Dry Mouth (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes